CLINICAL TRIAL: NCT06429059
Title: ROAR-DIGAP: A Widely Inclusive, Largely Virtual Pilot Trial Utilizing DIGAP (Deep Integrated Genomics Analysis Platform) To Personalize Treatments
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Temple University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00114385
Record Dates: First submitted 2024-04-09; First posted 2024-05-24 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-05

CONDITIONS: Amyotrophic Lateral Sclerosis ALS
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — astaxanthine; Protandim; Melatonin; mitoquinone

STUDY DESIGN:
Intervention Model Description: At month 3, DIGAP classification will be revealed to each participant and based on this, they will receive 1 of 4 treatments. They will take their assigned treatment for 6 months.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Neuroinflammation (Experimental): Study participants in this category are expected to have inflammation in their brains and spinal cords.
  Interventions: Drug: Astaxanthin
- Oxidative Stress (Experimental): Study participants in this category are expected to have too many damaging "free radical" chemicals in their brains and spinal cords.
  Interventions: Drug: Protandim
- Impaired Autophagy and Axonal Transport (Experimental): Study participants in this category are expected to have motor neurons that have trouble transporting materials up and down their length, and/or trouble with the turnover of damaged proteins and intracellular structures.
  Interventions: Drug: Melatonin
- Mitochondrial Dysfunction (Experimental): Study participants in this category are expected to have motor neurons that are unable to produce normal amounts of energy.
  Interventions: Drug: MitoQ

INTERVENTIONS:
Drug: Astaxanthin — Astaxanthin is a red-orange natural pigment belonging to a group of carotenoids called xanthophylls. In nature, astaxanthin is synthesized by microalgae and phytoplankton and biomagnifies in higher marine animals through the food chain. Natural astaxanthin is available as capsules, soft gels, tablets, powders, biomass, creams, energy drinks, oils and extracts and often contains other carotenoids. The compound is available as a United States Pharmacopeia (USP) verified supplement which ensures federally recognized standards for quality and purity (https://www.quality-supplements.org/verified-products/verified-products-listings).
  Arms: Neuroinflammation
Drug: Protandim — Protandim is an oral tablet derived from five different plants: Silybum marianum (milk thistle), Withania somnifera (Ashwagandha), Camellia sinensis (green tea), Curcuma longa (turmeric) and Bacopa monniera.
  Arms: Oxidative Stress
Drug: Melatonin — Melatonin is a hormone that has long been known to play a role in regulating sleep. Melatonin supplements are commonly used to treat insomnia, but in recent years, melatonin has been found to play a wider role in human physiology including the potential regulation of autophagy.
  Arms: Impaired Autophagy and Axonal Transport
Drug: MitoQ — The active ingredient in MitoQ is ubiquinone, the same as found in coenzyme Q10 and idebenone. However, the ubiquinone in MitoQ is attached to a positively charged, lipophilic molecule called TPP (triphenyl phosphonium), which allows it to selectively accumulate in mitochondria. This makes it more potent than untargeted ubiquinone analogs at protecting mitochondria in cultured cells. It can be administered orally and, at least in animals, can cross the blood brain barrier and accumulate in brain mitochondria.
  Arms: Mitochondrial Dysfunction

SUMMARY:
GenieUs developed an analysis platform that will be tested to separate study participants with ALS into four categories based on blood work. These general categories are neuroinflammation, oxidative stress, impaired autophagy & axonal transport, and mitochondrial dysfunction. Once a disease category is established, participants in this study will receive one of four individualized supplements for 6 months and we will determine whether these are slowing ALS progression: Astaxanthin will be given for the category of neuroinflammation, Protandim for oxidative stress, Melatonin for impaired autophagy and MitoQ for mitochondrial dysfunction. During the first 3 months, participants will have routine monitoring and in months 3 through 9 they will receive the assigned supplement.

DETAILED DESCRIPTION:
This will be a widely inclusive, largely remote/virtual, two-center, open-label pilot trial utilizing 50 participants as their own controls. Following informed consent and screening, participants will provide demographics, disease characteristics, co-morbidities, and concomitant medications. They will have a baseline ALSFRS-R score obtained and blood will be drawn for DIGAP classification, PBMCs (which will be used to generate iPSCs from which motor neurons and/or microglia can be generated), baseline mechanistic biomarkers and baseline neurofilament light chain. A urine pregnancy test will be obtained for pre-menopausal females who have not had one by their own doctor in the past 7 days. Each month after that, they will be contacted by phone by study coordinators to review adverse events, new co-morbidities, and concomitant medications, and to generate a new ALSFRS-R score. At month 3, DIGAP classification will be revealed to each participant and based on this, they will receive 1 of 4 treatments. They will take their assigned treatment for 6 months. At months 3, 5 and 9 they will be asked to return for in person blood draws for repeat mechanistic biomarkers and neurofilament light chain measurements. All of the described blood tests and investigational treatments are being performed exclusively for research purposes.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged at least 18 years.
2. Sporadic or familial ALS diagnosed as per Gold Coast Criteria.
3. Patient is able to understand and express informed consent (in the opinion of the site investigator).
4. Patient is able to read and write English.
5. Patient is expected to survive for the duration of the trial.
6. Able to swallow tablets at enrollment and expected to be able to swallow tablets for the duration of the trial.
7. Women must not be pregnant (will have evidence of a negative pregnancy test obtained by study team at baseline, or by local physician within past 7 days or be post-menopausal)
8. Women must not be able to become pregnant (e.g., post-menopausal, surgically sterile, or using adequate birth control methods) for the duration of the study and three months after study completion. Adequate contraception includes abstinence, hormonal contraception (oral contraception, implanted contraception, injected contraception, or other hormonal contraception, for example patch or contraceptive ring), intrauterine device (IUD) in place for ≥ 3 months, barrier method in conjunction with spermicide, or another adequate method.

Exclusion Criteria:

1. Actively or recently (within past 30 days) participating in another intervention trial.
2. Currently or recently (within 30 days) taking any of the 4 investigational treatments being used in this trial.
3. Prior side effects from any of the 4 investigational treatments being used in this trial.
4. Patient has a medical or psychiatric illness that could in the investigator's opinion interfere with the patient's ability to participate in this study.
5. Pregnant women or women currently breastfeeding.
6. Life expectancy shorter than the duration of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-06-12 (Actual); Primary Completion 2025-05-22 (Actual); Study Completion 2025-06-24 (Actual)

PRIMARY OUTCOMES:
ALS Functional Rating Scale, Revised (ALSFRS-R) | baseline and at each of the subsequent 9 telephone or in person visits (approximately 9 months)
  A quickly administered (five minute) ordinal rating scale (ratings 0-4) used to determine patients' assessments of their capability and independence in 12 functional activities. All 12 activities are relevant to people living with ALS.The ALSFRS-R declines linearly with time over a wide range during the course of ALS and it has been validated for telephone use.

SECONDARY OUTCOMES:
Neurofilament Light Chain levels | baseline, month 3, month 5 (2 months into treatment) and month 9 (6 months into treatment)
  They are neuron-specific components of the cytoskeleton. They exist in heavy, medium, and light chain forms. Neurofilament light chain levels are elevated in the spinal fluid and the blood of patients with ALS and other neurodegenerative diseases, and higher levels predict more severe disease progression. These levels rise dramatically when asymptomatic carriers of ALS-causing genetic mutations begin to convert to an ALS phenotype.
Neuroinflammation measured by C-reactive protein (CRP) | baseline, 3 months, 5 months and 9 months
  Used to measure neuroinflammation. These are known to be abnormal in patients with ALS, their levels correlate with disease progression and they can be altered by drugs in trials.
Neuroinflammation measured by monocyte chemoattractant protein-1 (MCP-1) | baseline, 3 months, 5 months and 9 months
  Used to measure neuroinflammation. These are known to be abnormal in patients with ALS, their levels correlate with disease progression and they can be altered by drugs in trials.
Neuroinflammation measured by chitotriosidase (CHIT1) | baseline, 3 months, 5 months and 9 months
  Used to measure neuroinflammation. These are known to be abnormal in patients with ALS, their levels correlate with disease progression and they can be altered by drugs in trials.
Oxidative stress measured by total antioxidant capacity (TAC) | baseline, 3 months, 5 months and 9 months
  Used to measure oxidative stress.
Oxidative stress measured by uric acid levels. | baseline, 3 months, 5 months and 9 months
  Uric acid is an antioxidant and levels of uric acid have been reported to be lower in ALS subjects and correlated with progression. It has also been shown to be responsive to treatments in trials
Impaired autophagy measured by Beclin-1 | baseline, 3 months, 5 months and 9 months
  To measure impaired autophagy, we will use Beclin-1. This highly conserved eukaryotic protein has a major regulatory role in autophagy. It is a component of the phosphatidylinositol-3-kinase (PI3K) complex which mediates vesicle-trafficking thereby inducing autophagy. Beclin-1 dysfunction has been implicated in many disorders, including cancer and neurodegenerative diseases
Mitochondrial dysfunction measured by lactate. | baseline, 3 months, 5 months and 9 months
  Compromised mitochondrial oxidative phosphorylation shifts the cellular bioenergetic system to anaerobic respiration and increases the level of lactate. Lactate has been used as a biomarker for mitochondrial disease in many previous studies.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Duke University Medical Center, Durham, North Carolina
  - Temple University, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No